CLINICAL TRIAL: NCT02815176
Title: Analysis of Plasminogen Activator Inhibitor-1 Level in Chronic Serous Chorioretinopathy and Polypoidal Choroidal Vasculopathy
Brief Title: Angiographic Characteristics of CSC, PCV Patients and Thrombotic Bio-markers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-02-109
Record Dates: First submitted 2016-06-13; First posted 2016-06-28 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Central Serous Chorioretinopathy; Polypoidal Choroidal Vasculopathy
Keywords: Plasminogen activator inhibitor-1; Wide angle fluorescein angiography; Choroid
MeSH Terms: conditions — Central Serous Chorioretinopathy; Polypoidal Choroidal Vasculopathy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples including DNA will be retained to perform the genotyping analysis of PAI-1 SNP.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Central serous chorioretinopathy: De novo eligible CSC patients will be allocated in this group. Blood sampling, fluorescein angiography, indocyanine green angiography will be performed within a week after initial diagnosis.
  Interventions: Other: Blood sampling
- Polypoidal choroidal vasculopathy: De novo eligible PCV patients will be allocated in this group. Blood sampling, fluorescein angiography, indocyanine green angiography will be performed within a week after initial diagnosis.
  Interventions: Other: Blood sampling
- Epiretinal membrane: Idiopathic ERM patients will be allocated in this group. Blood sampling, fluorescein angiography, indocyanine green angiography will be performed within a week after initial diagnosis.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Sampling the blood including DNA to investigate the thrombotic profile

SUMMARY:
Thrombotic biomarkers and angiographic characteristics were compared among the de novo patients of central serous chorioretinopathy (CSC), polypoidal choroidal vasculopathy (PCV) and the control.

ELIGIBILITY:
Inclusion Criteria:

* CSC

  * neurosensory detachment in optical coherence tomography (OCT)
  * focal leakage in fluorescein angiography (FAG) and/or late choroidal hyperpermeability in indocyanine green angiography (ICGA)
* PCV

  * subretinal and/or sub-retinal pigment epithelial fluid in OCT
  * branching vascular network and/or polyps in ICGA
* Control

  * epiretinal membrane (ERM)
  * without underlying systemic, ophthalmic disease other than ERM

Exclusion Criteria:

* Previous history of using steroid (oral, topical)
* Previous history of CSC/PCV
* Previous history or evidence of intraocular inflammation including uveitis
* Co-existing retinal or choroidal diseases
* History of allergic reaction to fluorescein or indocyanine green dye
* Underlying systemic conditions that could affect the thrombotic profiles (e.g. diabetes, hypertension, metabolic syndrome, coronary artery disease, cerebrovascular diseases, stroke, chronic renal failure, current smoker, pregnancy, sleep disorder)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: De novo patients with active CSC and PCV.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Serum Fibrinogen in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum Fibrinogen (mg/dl)
Serum Factor VIII activity in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum Factor VIII activity (%)
Serum Plasminogen activity in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum Plasminogen activity (%)
Serum D-dimer in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum D-dimer (μg/mL(FEU))
Serum Fibrin degradation product in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum Fibrin degradation product (μg/mL)
Serum PAI-1 antigen in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum PAI-1 (plasminogen activator inhibitor-1) antigen (ng/mL)
Serum PAI-1 SNP genotyping in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Serum PAI-1 SNP(single nucleotide polymorphism) genotyping

SECONDARY OUTCOMES:
Characteristics of fluorescein angiography in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Numbers of leaking points of fluorescein dye in fluorescein angiography
Characteristics of indocyanine green angiography in active PCV and CSC patients | Less than 1 week after initial diagnosis
  Numbers of hyperfluorescent spots in indocyanine green angiography

CONTACTS AND LOCATIONS:
Overall Officials: Kunho Bae, MD, Principal Investigator — Department of ophthalmology, Samsung medical center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No